CLINICAL TRIAL: NCT05598723
Title: A Randomized, Double-Blind Study on the Effect of OnabotulinumtoxinA (BOTOX®) vs. IncobotulinumtoxinA (XEOMIN®) Botulinum Toxin in Adults With Chronic Migraine
Brief Title: BOTOX® vs. XEOMIN® for Chronic Migraine
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Naval Medical Center Camp Lejeune (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NMCCL.2022.0029
Record Dates: First submitted 2022-10-25; First posted 2022-10-28 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2024-12

CONDITIONS: Chronic Migraine
Keywords: Botox; Xeomin; onabotulinumtoxinA; incobotulinumtoxinA; Botulinum Toxin; refrigeration; HIT-6
MeSH Terms: interventions — incobotulinumtoxinA; Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: A randomized, double blind, prospective, parallel-group study (non-inferiority trial)
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- OnabotulinumtoxinA (BOTOX®) (Active Comparator): OnabotulinumtoxinA (BOTOX®) Group: Administration consists of 31 injections (5 onabotulinumtoxinA (BOTOX®) units per injection, for a total of 155units) in the head and neck at two time points (12 weeks apart). Injection sites include the forehead, temples, back of the head, upper neck, and the junction of the shoulder and the neck. A very small (e.g., 30-gauge), very sharp needle will be used to perform the injections.
  Interventions: Drug: OnabotulinumtoxinA (BOTOX®)
- IncobotulinumtoxinA (XEOMIN®) (Experimental): IncobotulinumtoxinA (XEOMIN®) Group: Administration consists of 31 injections (5 incobotulinumtoxinA (XEOMIN®) units per injection, for a total of 155 units) in the head and neck at two time points (12 weeks apart). Injection sites include the forehead, temples, back of the head, upper neck, and the junction of the shoulder and the neck. A very small (e.g., 30-gauge), very sharp needle will be used to perform the injections.
  Interventions: Drug: IncobotulinumtoxinA (XEOMIN®)

INTERVENTIONS:
Drug: IncobotulinumtoxinA (XEOMIN®) — IncobotulinumtoxinA (XEOMIN®) is injected into specific targets at two different time points. Changes in chronic migraine frequency and duration are recorded and compared.
  Other Names: Xeomin
  Arms: IncobotulinumtoxinA (XEOMIN®)
Drug: OnabotulinumtoxinA (BOTOX®) — OnabotulinumtoxinA (BOTOX®) is injected into specific targets at two different time points. Changes in chronic migraine frequency and duration are recorded and compared.
  Other Names: Botox
  Arms: OnabotulinumtoxinA (BOTOX®)

SUMMARY:
Chronic migraine (CM) is a disabling disorder that sidelines active duty personnel and diminishes their quality of life. It affects 1.3% to 2.4% of the general population. These numbers increase in active duty personnel, especially those returning from deployment, as well as in veterans. Furthermore, these numbers are 4-5 times higher in military members who experienced at least one mild traumatic brain injury. CM leads to impaired cognition and poor decision-making. These impairments on critical active duty tasks could have a significant impact on task readiness and military performance. Therefore, CM presents a challenge for the "return to duty" mission. Currently, onabotulinumtoxinA is the only FDA-approved prophylactic treatment for CM; however, this treatment requires refrigeration, to which there is little access for the forward-deployed members who have limited access to adequate storage for this treatment. Therefore, it is imperative to identify a CM treatment that does not require refrigeration. Furthermore, in light of the ongoing COVID-19 pandemic and resulting international shortages in critical medication production and delivery, it is imperative to identify more than one treatment option for the management of CM. In this study, we will test the efficacy of incobotulinumtoxinA, a neurotoxin that, unlike onabotulinumtoxinA, does not require refrigeration, but is an effective off-label alternative for the treatment of migraine. OnabotulinumtoxinA and incobotulinumtoxinA are comparable in strength, with a conversion ratio of 1:1.

DETAILED DESCRIPTION:
One hundred and twenty-eight male and female active duty personnel, adult dependent and retiree patients from the Navy Medical Center at Camp Lejeune who meet the International Classification of Headache Disorders 3rd Edition (ICHD-3) criteria of ≥15 headache days per month lasting 4 hours or longer will participate in the trial. Subjects will be group-allocated randomly, 64 to onabotulinumtoxinA and 64 to incobotulinumtoxinA. Injections of either treatment will occur twice, 12 weeks apart, in the head and neck regions. The primary treatment efficacy measurement will be the mean change in headache days 12 to 24 weeks post-treatment. Participants will complete an electronic diary to report headache days, their severity, and adverse effects or unforeseen events. A baseline will be established four weeks prior to the first botulinumtoxinA (Botox or Xeomin) administration using the number of headache days and two questionnaires, Headache Impact Test-6 (HIT-6) and the Migraine Specific Quality (MSQ) Questionnaire, which assess headache impact and Health-Related Quality of Life (HRQOL), respectively. These questionnaires will also be administered at weeks 12 and 24 of the study. The baseline, 12-, and 24-week analysis will be performed using a time vs. treatment repeated measures analysis of variance for headache days. Secondary outcomes (total scores of both the HIT-6 and MSQ) will be analyzed similarly.

ELIGIBILITY:
Inclusion Criteria:

* Between ages of 18-89
* 15 or more headaches days experienced per month lasting 4 hours or longer
* Department of Defense (DoD) Beneficiary/TriCare Eligible
* Failure, contraindication or intolerance to two migraine medications from two different classes.
* Able to provide informed consent and be able to read and write English.
* Able to read, comprehend, and complete the assessment and diary
* Women must provide a negative urine pregnancy test

Exclusion Criteria:

* Currently pregnant, breastfeeding, or planning to become pregnant
* Allergic to botulinum toxin or to any of the ingredients of the medication
* Has myasthenia gravis, amyotrophic lateral sclerosis, or Eaton Lambert syndrome, mitochondrial disease, fibromyalgia, any temporomandibular disfunction, or any other significant disease that might interfere with neuromuscular function.
* Uncontrolled epilepsy defined as more than 1 generalized seizure in any month within the 3 months prior to the day 0 visit
* Those on oral anticoagulation
* Previous botulinum toxin treatment on the cephalic/upper lumbar region within 6 months for any indication
* Localized infections on face, neck or on antibiotics for areas in this region
* Unable to attend study follow up visits for any reason (i.e. Training, deployment, or PCS)
* Use of any prophylactic headache medication between -4 weeks and week 0 visits
* Any person taking chronic pain medication for a chronic indication
* Any diagnosed psychiatric condition which would prohibit a participant from completing the trial in its totality.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2023-02-24 (Actual); Primary Completion 2026-02-24 (Estimated); Study Completion 2026-08-24 (Estimated)

PRIMARY OUTCOMES:
Headache days per month | 24 weeks + Baseline
  To compare the difference in headache days per month (incobotulinumtoxinA (XEOMIN®) relative to onabotulinumtoxinA (BOTOX®)) at the end of treatment period (24 weeks).

SECONDARY OUTCOMES:
Differences in headache impact | 24 weeks vs. Baseline
  Assessed using the Headache Impact Test-6 (HIT-6): mean change from baseline will be reported. HIT-6 score ranges between 36 and 78, with larger scores reflecting greater impact.
Differences in Health-Related Quality of Life | 24 weeks vs. Baseline
  Assessed using the Migraine Specific Quality (MSQ) Questionnaire: mean change from baseline will be reported. MSQ score ranges between 0-100 scale, with higher scores signifying better health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline S Buckley, PharmD, Principal Investigator — Naval Medical Center Camp Lejeune
Locations (1):
- Naval Medical Center Camp Lejeune, Jacksonville, North Carolina, United States

REFERENCES:
- [Background] Burstein R, Noseda R, Borsook D. Migraine: multiple processes, complex pathophysiology. J Neurosci. 2015 Apr 29;35(17):6619-29. doi: 10.1523/JNEUROSCI.0373-15.2015. PMID 25926442
- [Background] Sandrini G, De Icco R, Tassorelli C, Smania N, Tamburin S. Botulinum neurotoxin type A for the treatment of pain: not just in migraine and trigeminal neuralgia. J Headache Pain. 2017 Dec;18(1):38. doi: 10.1186/s10194-017-0744-z. Epub 2017 Mar 21. PMID 28324318
- [Background] May A, Schulte LH. Chronic migraine: risk factors, mechanisms and treatment. Nat Rev Neurol. 2016 Aug;12(8):455-64. doi: 10.1038/nrneurol.2016.93. Epub 2016 Jul 8. PMID 27389092
- [Background] Schwedt TJ. Chronic migraine. BMJ. 2014 Mar 24;348:g1416. doi: 10.1136/bmj.g1416. PMID 24662044
- [Background] Headache Classification Committee of the International Headache Society (IHS). The International Classification of Headache Disorders, 3rd edition (beta version). Cephalalgia. 2013 Jul;33(9):629-808. doi: 10.1177/0333102413485658. No abstract available. PMID 23771276
- [Background] Do TP, Hvedstrup J, Schytz HW. Botulinum toxin: A review of the mode of action in migraine. Acta Neurol Scand. 2018 May;137(5):442-451. doi: 10.1111/ane.12906. Epub 2018 Feb 6. PMID 29405250
- [Background] Carruthers A, Carruthers J. Botulinum toxin products overview. Skin Therapy Lett. 2008 Jul-Aug;13(6):1-4. PMID 18806905
- [Background] Frevert J, Dressler D. Complexing proteins in botulinum toxin type A drugs: a help or a hindrance? Biologics. 2010 Dec 9;4:325-32. doi: 10.2147/BTT.S14902. PMID 21209727
- [Background] Aurora SK, Dodick DW, Turkel CC, DeGryse RE, Silberstein SD, Lipton RB, Diener HC, Brin MF; PREEMPT 1 Chronic Migraine Study Group. OnabotulinumtoxinA for treatment of chronic migraine: results from the double-blind, randomized, placebo-controlled phase of the PREEMPT 1 trial. Cephalalgia. 2010 Jul;30(7):793-803. doi: 10.1177/0333102410364676. Epub 2010 Mar 17. PMID 20647170
- [Background] Diener HC, Dodick DW, Aurora SK, Turkel CC, DeGryse RE, Lipton RB, Silberstein SD, Brin MF; PREEMPT 2 Chronic Migraine Study Group. OnabotulinumtoxinA for treatment of chronic migraine: results from the double-blind, randomized, placebo-controlled phase of the PREEMPT 2 trial. Cephalalgia. 2010 Jul;30(7):804-14. doi: 10.1177/0333102410364677. Epub 2010 Mar 17. PMID 20647171
- [Background] Rendas-Baum R, Bloudek LM, Maglinte GA, Varon SF. The psychometric properties of the Migraine-Specific Quality of Life Questionnaire version 2.1 (MSQ) in chronic migraine patients. Qual Life Res. 2013 Jun;22(5):1123-33. doi: 10.1007/s11136-012-0230-7. Epub 2012 Jul 15. PMID 22797868
- [Background] Ion I, Renard D, Le Floch A, De Verdal M, Bouly S, Wacongne A, Lozza A, Castelnovo G. Monocentric Prospective Study into the Sustained Effect of Incobotulinumtoxin A (XEOMIN(R)) Botulinum Toxin in Chronic Refractory Migraine. Toxins (Basel). 2018 Jun 1;10(6):221. doi: 10.3390/toxins10060221. PMID 29857565
- [Background] Kwong WJ, Pathak DS. Validation of the eleven-point pain scale in the measurement of migraine headache pain. Cephalalgia. 2007 Apr;27(4):336-42. doi: 10.1111/j.1468-2982.2007.01283.x. PMID 17376110
- [Background] Bagley CL, Rendas-Baum R, Maglinte GA, Yang M, Varon SF, Lee J, Kosinski M. Validating Migraine-Specific Quality of Life Questionnaire v2.1 in episodic and chronic migraine. Headache. 2012 Mar;52(3):409-21. doi: 10.1111/j.1526-4610.2011.01997.x. Epub 2011 Sep 19. PMID 21929662
- [Background] Wilderman I, Tallarigo D, Pugacheva-Zingerman O. A Qualitative Study to Explore Patient Perspectives of Prophylactic Treatment with OnabotulinumtoxinA for Chronic Migraine. Pain Ther. 2021 Dec;10(2):1523-1536. doi: 10.1007/s40122-021-00316-2. Epub 2021 Sep 14. PMID 34523107
- [Background] Stark C, Stark R, Limberg N, Rodrigues J, Cordato D, Schwartz R, Jukic R. Real-world effectiveness of onabotulinumtoxinA treatment for the prevention of headaches in adults with chronic migraine in Australia: a retrospective study. J Headache Pain. 2019 Jul 15;20(1):81. doi: 10.1186/s10194-019-1030-z. PMID 31307383
- [Background] Kawata AK, Shah N, Poon JL, Shaffer S, Sapra S, Wilcox TK, Shah S, Tepper SJ, Dodick DW, Lipton RB. Understanding the migraine treatment landscape prior to the introduction of calcitonin gene-related peptide inhibitors: Results from the Assessment of TolerabiliTy and Effectiveness in MigrAINe Patients using Preventive Treatment (ATTAIN) study. Headache. 2021 Mar;61(3):438-454. doi: 10.1111/head.14053. Epub 2021 Feb 16. PMID 33594686
- [Background] Kreidler SM, Muller KE, Grunwald GK, Ringham BM, Coker-Dukowitz ZT, Sakhadeo UR, Baron AE, Glueck DH. GLIMMPSE: Online Power Computation for Linear Models with and without a Baseline Covariate. J Stat Softw. 2013 Sep;54(10):i10. doi: 10.18637/jss.v054.i10. PMID 24403868
- [Background] Yiannakopoulou E. Serious and long-term adverse events associated with the therapeutic and cosmetic use of botulinum toxin. Pharmacology. 2015;95(1-2):65-9. doi: 10.1159/000370245. Epub 2015 Jan 21. PMID 25613637
- [Background] Kessler KR, Skutta M, Benecke R. Long-term treatment of cervical dystonia with botulinum toxin A: efficacy, safety, and antibody frequency. German Dystonia Study Group. J Neurol. 1999 Apr;246(4):265-74. doi: 10.1007/s004150050345. PMID 10367694
- [Background] Fisher CM. Late-life migraine accompaniments--further experience. Stroke. 1986 Sep-Oct;17(5):1033-42. doi: 10.1161/01.str.17.5.1033. PMID 3532432
- [Background] Naumann M, Jankovic J. Safety of botulinum toxin type A: a systematic review and meta-analysis. Curr Med Res Opin. 2004 Jul;20(7):981-90. doi: 10.1185/030079904125003962. PMID 15265242